CLINICAL TRIAL: NCT00857883
Title: A First-Time-In-Human, Three-Part, Placebo-Controlled, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK1521498 in Healthy Subjects
Brief Title: A First-Time-In-Human Study in Healthy Subjects
Acronym: FTIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111314
Record Dates: First submitted 2009-02-24; First posted 2009-03-09 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: Obesity; Food Effect; Pharmacokinetics; First-Time-In-Humans; Pharmacodynamics; Healthy Volunteers
MeSH Terms: conditions — Obesity | interventions — N-((3,5-difluoro-3'-(1H-1,2,4-triazol-3-yl)-4-biphenylyl)methyl)-2,3-dihydro-1H-inden-2-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Placebo Comparator): Part A: This part of the study will start with a very low dose of study drug, which will then be gradually increased in subsequent doses. This is known as dose-rising and is the way to assess safety and tolerability (i.e. possible presence of any side effects that make taking the drug unpleasant) of increasing doses of the study drug. Effects will be compared to those seen when a placebo is taken. Up to 4 groups of 6-9 healthy male or female volunteers will be enrolled.
  Interventions: Drug: GSK1521498 or placebo
- Part B (Active Comparator): Part B: A dose selected from Part A that was well tolerated will be used to check if there is a difference in the pharmacokinetics (blood levels) of the study drug when taken without food in liquid form, or as a capsule, or as a capsule together with a high fat meal to assess the effect of food. One group of 12 healthy male or female volunteers will be enrolled.
  Interventions: Drug: GSK1521498 or placebo
- Part C (Placebo Comparator): Part C: A well tolerated dose selected from Parts A & B will be used to test whether the drug has an effect on individual preferences for sugary and high fat food, when compared to placebo. Up to 32 healthy overweight male volunteers will be enrolled.
  Interventions: Drug: GSK1521498 or placebo

INTERVENTIONS:
Drug: GSK1521498 or placebo — GSK1521498 is a mu-opioid receptor inverse agonist

SUMMARY:
This is a first-time-in-human study. The overall purpose of the study is to assess whether the drug is safe and well tolerated after single, increasing doses. The blood levels of the drug after different doses will be measured and the effect of the drug on pleasurable eating behaviour will be assessed.

DETAILED DESCRIPTION:
The human body naturally produces substances known as opioids and the pleasurable (or hedonic) response to eating highly sugary or fatty foods is increased by opioids. The drug to be tested in this study attaches to specific binding sites in the brain, known as mu-opioid receptors. This may stop the natural effect of opioids and therefore reduce the pleasurable response to food. We predict that this in turn may help patients with obesity to lose weight more effectively. The study is divided into three parts:

Part A: This part of the study will start with a very low dose of study drug, which will then be gradually increased in subesquent doses. This is known as dose-rising and is the way to assess safety and tolerability (any side effects that make taking the drug unpleasant). Effects will be compared to those seen when a placebo (a "dummy" drug) is taken. Up to 4 groups of 6-9 healthy male or female volunteers will be enrolled in this part of the study.

Part B: A dose selected from Part A that was well tolerated will be used to check if there is a difference in the blood levels of the study drug when taken without food in liquid form, without food as a capsule, or with a high fat meal as a capsule. One group of 12 healthy male or female volunteers will be enrolled in this part of the study.

Part C: A well tolerated dose selected from Parts A & B will be used to test whether the drug has an effect on preferences for sugary and high fat food, when compared to placebo. Up to 32 healthy overweight male volunteers will be enrolled in this part of the study.

ELIGIBILITY:
Inclusion Criteria:

- Part A and Part B: Healthy male or female subject as determined by a responsible physician, based on a medical evaluation including history, physical examination, vital signs, laboratory tests and cardiac monitoring. Male subjects must agree to use one of the contraception methods listed in Section 8 from dosing until 84 days after the last dosing session.

Female subjects must be of non-childbearing potential including pre-menopausal women with documented (medical report verification) hysterectomy, tubal ligation, or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

Part C: Only healthy male subjects will be enrolled (females not included due to the potential influence of the menstrual cycle on eating behaviour). Male subjects must agree to use one of the contraception methods listed in Section 8 from dosing until 84 days after the last dosing session.

* Between 18 and 50 years of age, inclusive, at the time of signing and dating the informed consent form.
* Body weight > 45 kg and BMI within the range 20 - 30 kg/m2 (inclusive) for Part A and B and a BMI within the range 25 - 35 kg/m2 (inclusive) for Part C.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* A history of uncorrected thyroid dysfunction or an abnormal thyroid function test assessed by TSH at screening
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to 8g of alcohol, a half-pint (~240 mL) of beer or 1 (25 ml) measure of spirits or 1 glass (125 ml) of wine.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Has a history of any gastrointestinal or hepatic conditions that could affect absorption of the investigational product.
* Has QTc at screening > 450 msec. Note that if the initial QTc value is prolonged, the ECG should be repeated two more times (with 5 minutes between ECG readings) and the average of the 3 QTc values used to determine eligibility.
* Has clinically significant rhythm abnormalities identified during 24-hour screening Holter assessment.
* Systolic BP outside the range 85 to 160 mmHg, diastolic BP outside the range 45 to 100 mmHg, and/or heart rate outside the range 40 to 110 bpm.
* Self-administered Beck Depression Inventory II scale total score greater than nine. Suicide question score greater than zero.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months before or after the study.
* Unwilling to abstain from:
* Consumption of caffeine- or xanthine containing products for 24 hours prior to dosing until the post-dose assessment at each treatment level.
* Use of illicit drugs
* Alcohol for 48 hours prior to dosing until final post-dose assessment at each treatment level
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the dose of study medication until collection of the final pharmacokinetic blood sample.
* Vegans and milk intolerance as reported by the subject (Part C only)
* Unwillingness or inability to follow the procedures outlined in the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-01 (Actual)

PRIMARY OUTCOMES:
Safety: adverse events, changes in clinical chemistry, haematology, urine parameters, blood pressure, heart rate, ECG, Bond & Lader visual Analog Scale, Profile of Mood States | 19 weeks
Tolerability: adverse events, changes in clinical chemistry, haematology, urine parameters, blood pressure, heart rate, ECG, Bond & Lader visual Analog Scale, Profile of Mood States | 19 weeks
Pharmacokinetic parameters | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post dose administrations

SECONDARY OUTCOMES:
Bioavailability of liquid form of drug and capsule and effect of food on the capsule | Approx 4 weeks
Pharmacodynamics - response to sweet and high fat foods before and after drug administration | Approx 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 111314 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111314?search=study&study_ids=111314#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register